CLINICAL TRIAL: NCT01229891
Title: Comparison of Efficacy of Vitamin D and Vitamin D-calcium Fortified Yogurt Drink on Glycemic, Metabolic, Inflammatory, Immunity and Oxidative Stress Markers in Type 2 Diabetes
Brief Title: Comparison of Efficacy of Vitamin D and Vitamin D-calcium Fortified Yogurt Drink in Diabetic Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Nutrition and Food Technology Institute (Other)
Responsible Party: Principal Investigator, Tirang R. Neyestani, associate professor, National Nutrition and Food Technology Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 11024
Record Dates: First submitted 2010-10-27; First posted 2010-10-28 (Estimated); Results first posted 2012-01-16 (Estimated); Last update posted 2012-01-16 (Estimated); Status verified 2011-12

CONDITIONS: Type 2 Diabetes
Keywords: vitamin D fortification; yogurt drink; type 2 diabetes; efficacy
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Plain yogurt drink (Placebo Comparator): daily intake of two bottle (250 mL) plain yogurt drink
  Interventions: Dietary Supplement: plain yogurt drink
- vitamin D-fortified yogurt drink (Experimental): daily intake of two bottle yogurt drink fortified with 500 IU vitamin D/250 mL
  Interventions: Dietary Supplement: vitamin D fortified yogurt drink
- vitamin D-calcium yogurt drink (Experimental): daily intake of two bottle of yogurt drink fortified with 500 IU vitamin D and 250 mg calcium/250 mL
  Interventions: Dietary Supplement: vitamin D-calcium yogurt drink

INTERVENTIONS:
Dietary Supplement: plain yogurt drink — daily intake of two bottle of plain yogurt drink
  Other Names: PY
  Arms: Plain yogurt drink
Dietary Supplement: vitamin D fortified yogurt drink — daily intake of two bottle of yogurt drink fortified with 500 IU vitamin D/250 mL
  Other Names: DY
  Arms: vitamin D-fortified yogurt drink
Dietary Supplement: vitamin D-calcium yogurt drink — daily intake of two bottle of yogurt drink fortified with 500 IU vitamin D and 250 mg calcium/250 ml package
  Other Names: DCY
  Arms: vitamin D-calcium yogurt drink

SUMMARY:
The aim of this study is to evaluate the possible effects of daily intake of yogurt drink fortified with vitamin D alone or with vitamin D + calcium on some selected glycemic, metabolic, inflammatory and oxidative stress markers in patients with type 2 diabetes (T2DM).

DETAILED DESCRIPTION:
ninety diabetic patients will be selected. Patients who are receiving vitamin D, calcium or omega-3 supplements within the last three months will be excluded. Patients will be assigned randomly to one of the three intervention groups. 1. Plain yogurt drink 2. Vitamin D-fortified yogurt drink 3. Vitamin D-calcium fortified yogurt drink. Each patient will consume 2 servings of yogurt drink every day for 3 months with lunch and dinner. At the first and last visits, dietary and laboratory assessments will be performed for all patients. Primary outcomes are improvement in glycemic, inflammatory and immunity markers and secondary outcome is prevention of long-term diabetic complications.

ELIGIBILITY:
Inclusion Criteria:Age:

* 30 to 50 years,
* Fasting blood glucose ≥ 126 mg/dl

Exclusion Criteria:

* Receiving vitamin D or calcium or omega-3 supplements within the last three months,
* On any medication which could potentially influence vitamin D metabolism (notably estrogens, and calcitonin) within the last three months,
* Any other concomitant disease such as renal, hepatic, and other endocrinological disorders, and malignancies, which could influence vitamin D metabolism.
* Receiving insulin or any change in the type and/or dose of the current hypoglycemic medications

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2009-10; Primary Completion 2010-03 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tirang R. Neyestani, PhD, Study Chair — National Nutrition and Food Technology Research Institute

REFERENCES:
- [Derived] Nikooyeh B, Shariatzadeh N, Rismanchi M, Hollis BW, Neyestani TR. Daily intake of yogurt drink fortified either with vitamin D alone or in combination with added calcium causes a thyroid-independent increase of resting metabolic rate in adults with type 2 diabetes: a randomized, double-blind, clinical trial. Appl Physiol Nutr Metab. 2021 Nov;46(11):1363-1369. doi: 10.1139/apnm-2021-0248. Epub 2021 Jun 2. PMID 34077684
- [Derived] Heravifard S, Neyestani TR, Nikooyeh B, Alavi-Majd H, Houshiarrad A, Kalayi A, Shariatzadeh N, Zahedirad M, Tayebinejad N, Salekzamani S, Khalaji N, Gharavi A. Regular consumption of both vitamin D- and calcium- and vitamin D-fortified yogurt drink is equally accompanied by lowered blood lipoprotein (a) and elevated apoprotein A1 in subjects with type 2 diabetes: a randomized clinical trial. J Am Coll Nutr. 2013;32(1):26-30. doi: 10.1080/07315724.2013.767659. PMID 23875809
- [Derived] Neyestani TR, Nikooyeh B, Alavi-Majd H, Shariatzadeh N, Kalayi A, Tayebinejad N, Heravifard S, Salekzamani S, Zahedirad M. Improvement of vitamin D status via daily intake of fortified yogurt drink either with or without extra calcium ameliorates systemic inflammatory biomarkers, including adipokines, in the subjects with type 2 diabetes. J Clin Endocrinol Metab. 2012 Jun;97(6):2005-11. doi: 10.1210/jc.2011-3465. Epub 2012 Mar 22. PMID 22442277
- [Derived] Nikooyeh B, Neyestani TR, Farvid M, Alavi-Majd H, Houshiarrad A, Kalayi A, Shariatzadeh N, Gharavi A, Heravifard S, Tayebinejad N, Salekzamani S, Zahedirad M. Daily consumption of vitamin D- or vitamin D + calcium-fortified yogurt drink improved glycemic control in patients with type 2 diabetes: a randomized clinical trial. Am J Clin Nutr. 2011 Apr;93(4):764-71. doi: 10.3945/ajcn.110.007336. Epub 2011 Feb 2. PMID 21289226

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Plain Yogurt Drink | Vitamin D-fortified Yogurt Drink | Vitamin D-calcium Yogurt Drink
Started | 30 | 30 | 30
Completed | 30 | 30 | 30
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Plain Yogurt Drink | Vitamin D-fortified Yogurt Drink | Vitamin D-calcium Yogurt Drink | Total
Number analyzed (Participants) | 30 | 30 | 30 | 90
Age Continuous [Mean (Standard Deviation); unit: years] | 50.8 (6.6) | 51.4 (5.4) | 49.9 (6.2) | 50.7 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 16 | 9 | 43
  Male | 12 | 14 | 21 | 47
25-hydroxyvitamin D [Mean (Standard Deviation); unit: nmol/L] | 50 (26) | 47.5 (27) | 51.3 (43) | 48.8 (38.4)
Fasting serum glucose (FSG) [Mean (Standard Deviation); unit: mg/dL] — Fasting serum glucose concentration
  mg/dL | 187 (57.1) | 184.1 (63.8) | 184 (57.3) | 185 (58.8)
Insulin [Mean (Standard Deviation); unit: mU/L] — Fasting serum Insulin concentration
  mU/L | 7.7 (3.2) | 7.7 (4.6) | 7.6 (4.6) | 7.6 (4.1)
HbA1c [Mean (Standard Deviation); unit: percent] — Hemoglobin A1c
  percent | 7.5 (1.5) | 7.4 (1.8) | 7.8 (1.9) | 7.6 (1.7)
TG [Mean (Standard Deviation); unit: mg/dL] — serum triglyceride concentration
  mg/dL | 160.5 (100.7) | 155.4 (65.9) | 176.6 (91.0) | 164.2 (86.6)
Tchol [Mean (Standard Deviation); unit: mg/dL] — serum total cholesterol concentration
  mg/dL | 187.5 (43.3) | 177.5 (41.9) | 187.7 (46.6) | 182.4 (43.8)
LDL [Mean (Standard Deviation); unit: mg/dL] — serum low density lipoprotein concentration
  mg/dL | 88.6 (25.9) | 87.2 (25.1) | 90.2 (27.9) | 88.7 (26.0)
HDL [Mean (Standard Deviation); unit: mg/dL] — serum High density lipoprotein concentration
  mg/dL | 50.8 (8.2) | 46 (9.6) | 47.2 (9.4) | 48 (9.2)

OUTCOME MEASURES:

1. Primary Outcome: Serum 25-hydroxyvitamin D
Time Frame: 12-week
Measure: Mean (Standard Deviation); unit: nmol/L
Groups:
- Plain Yogurt Drink: 2 bottle plain yogurt drink per day
- Vitamin D-fortified Yogurt Drink: 2 bottle vitamin D-fortified yogurt drink per day
- Vitamin D-calcium Fortified Yogurt Drink: 2 bottle vitamin D-calcium-fortified yogurt drink per day
Arm/Group | Plain Yogurt Drink | Vitamin D-fortified Yogurt Drink | Vitamin D-calcium Fortified Yogurt Drink
Number analyzed (Participants) | 30 | 30 | 30
nmol/L | 45.6 (45.4) | 76.2 (28.4) | 78.4 (40.8)

2. Secondary Outcome: Fasting Serum Glucose (FSG)
Time Frame: 12-week
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Plain Yogurt Drink | Vitamin D-fortified Yogurt Drink | Vitamin D-calcium Fortified Yogurt Drink
Number analyzed (Participants) | 30 | 30 | 30
mg/dL | 203.3 (64.4) | 171.2 (59.2) | 174.3 (50)

3. Secondary Outcome: Insulin
Description: fasting serum insulin concentration
Time Frame: 12-week
Measure: Mean (Standard Deviation); unit: mU/L
Arm/Group | Plain Yogurt Drink | Vitamin D-fortified Yogurt Drink | Vitamin D-calcium Fortified Yogurt Drink
Number analyzed (Participants) | 30 | 30 | 30
mU/L | 10.8 (5.5) | 6.5 (3.3) | 6.4 (3.1)

4. Secondary Outcome: Hemoglobin A1c (HbA1c)
Time Frame: 12-week
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Plain Yogurt Drink | Vitamin D-fortified Yogurt Drink | Vitamin D-calcium Fortified Yogurt Drink
Number analyzed (Participants) | 30 | 30 | 30
percent | 8.7 (1.4) | 7 (2.3) | 7.8 (1.9)

5. Secondary Outcome: Serum Triglyceride (TG)
Time Frame: 12-week
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Plain Yogurt Drink | Vitamin D-fortified Yogurt Drink | Vitamin D-calcium Fortified Yogurt Drink
Number analyzed (Participants) | 30 | 30 | 30
mg/dL | 181.3 (91.8) | 155.2 (55.1) | 161.1 (64.3)

6. Secondary Outcome: Serum Total Cholesterol (Tchol)
Time Frame: 12-week
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Plain Yogurt Drink | Vitamin D-fortified Yogurt Drink | Vitamin D-calcium Fortified Yogurt Drink
Number analyzed (Participants) | 30 | 30 | 30
mg/dL | 197.3 (48.1) | 182.8 (43.0) | 178.5 (42.4)

7. Secondary Outcome: Serum Low Density Lipoprotein (LDL)
Time Frame: 12-week
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Plain Yogurt Drink | Vitamin D-fortified Yogurt Drink | Vitamin D-calcium Fortified Yogurt Drink
Number analyzed (Participants) | 30 | 30 | 30
mg/dL | 93.5 (24.9) | 91.1 (19.8) | 96.3 (27.8)

8. Secondary Outcome: Serum High Density Lipoprotein (HDL)
Time Frame: 12-week
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Plain Yogurt Drink | Vitamin D-fortified Yogurt Drink | Vitamin D-calcium Fortified Yogurt Drink
Number analyzed (Participants) | 30 | 30 | 30
mg/dL | 51.8 (9.6) | 46.1 (10) | 48 (6.8)

ADVERSE EVENTS:
Time Frame: during the intervention (12-week)
Arm/Group | Plain Yogurt Drink | Vitamin D-fortified Yogurt Drink | Vitamin D-calcium Yogurt Drink
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes